CLINICAL TRIAL: NCT07061405
Title: Impact of a Multidisciplinary Rehabilitation Program and Doado Application on the Functional Disability of Patients With Low Back Pain at Risk of Chronicization, Compared With a Monodisciplinary Rehabilitation Program and Doado Application.
Brief Title: Impact of a Multidisciplinary Rehabilitation Program Associated With the Doado Application in Lowback Pain Management
Acronym: REEDUCALGIE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REEDUCALGIE
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Lumbar Pain Syndrome
Keywords: rehabilitation; functional disability; multidisciplinary program; physiotherapy
MeSH Terms: conditions — Somatoform Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multidisciplinary management associated with mobile application Doado (Experimental): 10 half-day sessions, in a day hospital, for 2 weeks, 5 times a week (Monday to Friday), each comprising 3 workshops, with the following contributors: physiotherapist, doctor, nurse, occupational therapist, psychologist, dietician, Adapted Physical Activity (APA) teacher. This program is associated with the Doado mobile application.
  The Doado mobile application includes rehabilitation exercises and educational content, to be used at home by the patients.
  Interventions: Other: Multidisciplinary management associated with mobile application Doado
- Physiotherapy management alone associated with mobile application Doado (Active Comparator): 10 active functional re-education sessions (1 hour), 2 to 3 per week (sessions are therefore spread over approximately 4 to 5 weeks), based on muscle-strengthening exercises for the trunk and lower limbs, as well as stretching exercises for the back and lower limbs. This program is associated with the Doado mobile application.
  Interventions: Other: Physiotherapy management alone associated with mobile application Doado

INTERVENTIONS:
Other: Multidisciplinary management associated with mobile application Doado — multidisciplinary program including physiotherapists, rheumatologists, physical medicine and rehabilitation specialists, occupational physicians, psychologists, etc., associated with Doado mobile application
  Arms: Multidisciplinary management associated with mobile application Doado
Other: Physiotherapy management alone associated with mobile application Doado — monodisciplinary physiotherapy rehabilitation program consisting of active treatment with a physiotherapist associated with Doado mobile application
  Arms: Physiotherapy management alone associated with mobile application Doado

SUMMARY:
This study is aimed at patients consulting a physiotherapist for acute low-back pain at risk of becoming chronic.

The goal of this study is to compare two types of rehabilitation programs for these patients, on their functional disability at 3 months:

* A multidisciplinary program lasting two weeks, including physiotherapists, rheumatologists, physical medicine and rehabilitation specialists, occupational physicians, psychologists, etc.
* A monodisciplinary physiotherapy rehabilitation program consisting of active treatment with a physiotherapist, with 2 to 3 sessions per week for 4 to 5 weeks, based on muscle-strengthening exercises for the trunk and lower limbs and stretching exercises for the back and lower limbs.

Patients will be evaluated before treatment (baseline), and at 1, 3, 6 and 12 months to evaluate the following secondary outcomes: pain, absence of chronicity, evolution of functional disability, muscle endurance, flexibility, level of fear, apprehension and avoidance associated with low back pain over the time, return to work and to physical activities, painful relapses and analgesic treatment consumption.

ELIGIBILITY:
Inclusion Criteria:

Patient:

1. Suffering from acute common low back pain for less than 3 months at the time of the initial consultation
2. With a prescription for physiotherapy
3. Available for both programs
4. Aged between 20 and 55
5. Equipped with a smartphone compatible with the Doado application
6. Having been informed and having signed the free and informed consent form prior to any specific study procedure
7. Affiliated to a health insurance scheme

Exclusion Criteria:

Patient:

1. suffering from a first episode of acute common low back pain for less than one month at the time of the initial consultation
2. With a history of spinal surgery:

   1. For lumbar arthrodesis in the 12 months prior to inclusion
   2. For lumbar arthroplasty in the 6 months prior to inclusion
   3. For lumbar recalibration or lumbar disc herniation within 3 months of inclusion.
3. With suspected specific low-back pain
4. Suffering from radiculalgia of the lower limbs
5. Suffering from sensory-motor disorders of the lower limbs
6. Suffering from continuous low-back pain for at least 3 months
7. Have severely impaired physical and/or psychological health, which in the investigator's opinion may affect the participant's compliance with the study.
8. Participating in other interventional research
9. In a period of exclusion from other research still in progress at the time of inclusion.
10. Protected: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision.
11. Pregnant, breast-feeding or parturient.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Functional disability | baseline, 3 months
  Oswestry disability Index (ODI): 10 questions with 6 possible answers each, to assess the impact of the pain on several life habits and functionalities (walk, personal care, sitting position, etc.). The score is expressed as a percentage of handicap between 0 and 100%.

SECONDARY OUTCOMES:
Lumbar pain | baseline, one month, 3 months, 6 months, 12 months
  Mean patient lumbar pain on the last 7 days measured on a visual analog scale. It takes the form of a horizontal line with a qualifier at each end - "no pain (0)" on the left, "maximum imaginable pain (10)" on the right - onto which the patient draws a line (or positions a cursor on the online version), corresponding to the level of intensity of their pain.
  The result is the distance in mm between 0 and the line.
Lumbar pain chronicity | over 12 months of follow-up
  Presence of lumbar pain chronicity, defined by daily continuous pain during at least 12 weeks. This data will be collected from the start and end dates of each recurrence entered by the patient in the patient logbook.
Functional disability | Baseline, one month, 3 months, 6 months, 12 months
  Oswestry disabilty Index
Muscular endurance (Shirado-Ito test) | baseline, one month, 3 months
  The patient must remain as long as possible with the hips and knees bent at 90°, shoulder blades lifted, arms crossed over torso and hands resting on shoulders. The test result is the time, in seconds, that the patient remains in this position (for a maximum of 5 minutes), measured by the physiotherapist using a stopwatch.
Muscular endurance (hip bridge endurance) | baseline, one month, 3 months
  The patient lies on his or her back on a flat surface, knees bent and feet flat on the floor, positioned hip-width apart. Arms are crossed over the chest. The patient lifts his hips toward the ceiling, lifting his pelvis off the floor. When his shoulders are in line with his pelvis and knees, he stretches out his left leg, taking off the heel of the same leg so that there is alignment between shoulders, pelvis, knees and lifted foot. The stopwatch is then started.
  The patient holds this position for as long as possible, without letting the hips collapse or releasing the leg in the air. The result is timed in seconds, measured by the physiotherapist.
  The timer is stopped as soon as a change of at least 10 degrees in the alignment of the transverse or sagittal plane is visually detected by the physiotherapist.
  The test is done on both sides (left and right). The result is expressed in seconds.
Muscular endurance (Biering-Sorensen) | baseline, one month, 3 months
  The patient is positioned on a Roman lumbar extension chair, prone with trunk in the air, arms crossed over the chest. The pelvis rests on the support up to the level of the anterior superior iliac spines. The lower limbs and pelvis are supported by the wedges. The patient must keep the trunk horizontal for as long as possible (within 4 minutes). The result is measured in seconds by the physiotherapist.
Muscular endurance (Killy test) | baseline, one month, 3 months
  The patient simulates sitting on a chair, back and head pressed against the wall, hips and knees bent at 90° but not touching, hands touching the wall but not resting against it. The patient must hold the position for as long as possible. The result is timed in seconds, measured by the physiotherapist. The stopwatch is stopped as soon as : shoulders lift off the wall, the patient's pelvis moves up the wall, so that the thighs are no longer parallel to the floor, the hands rest on the thighs or on the wall (as this facilitates positioning).
Flexibility (finger-ground distance test) | baseline, one month, 3 months
  Standing with feet together, the patient slowly tilts the chest forward, uncoiling the back with arms outstretched, in an attempt to touch the ground with the fingers, without bending the knees. The result of the test is the distance between the fingertips and the ground, measured with a ruler (cm). If the patient manages to touch the ground with the fingers and could go beyond this distance, the value will be scored at 0.
Flexibility (knee extension angle test) | expressed in degrees of amplitude Time Frame : baseline, one month, 3 months
  The patient lies supine, while the physiotherapist flexes the hip and extends the knee. An inclinometer is placed on the patient's tibia to quantify amplitude. Alternatively, a goniometer can be used. The test is repeated on the opposite side. By comparing the right and left amplitudes, if the practitioner notes an angular amplitude deficit, this may reflect a hamstring amplitude deficit. The test result is expressed in degrees of amplitude.
Flexibility (hill-ischin procubitus measurement test) | baseline, one month, 3 months
  The patient lies prone (procubitus) on a flat, comfortable surface. Legs should be fully extended and parallel. A tape measure is placed so that one end is aligned with the heel of the foot (posterior part of the heel) and the other end is directed towards the ischium (pelvic bone). The patient bends the knee of one leg as far as it will go, while keeping the other leg fully extended.
  The test result is the distance between the heel of the extended leg and the ischium on the same side, measured in cm.
Fear, apprehension and avoidance related to low back pain (SBST questionnaire) | baseline, one month, 3 months, 6 months, 12 months
  Start Back Screening Tool (SBST) is a 9 items questionnaire which identifies the presence of potentially modifiable physical and psychological indicators, persistent and disabling symptoms among patients suffering from low back pain. The result is a score between 0 and 9.
Fear, apprehension and avoidance related to low back pain (FABQ questionnaire) | baseline, one month, 3 months, 6 months, 12 months
  Fear Avoidance Belief Questionnaire (FABQ) is an assessment tool used in low back pain patients to measure patients' beliefs and attitudes about pain and physical activity, particularly in the context of musculoskeletal pain. It assesses how fear of pain may influence physical activity avoidance behavior. There are two subscales in the FABQ: the work subscale (FABQw) with 7 questions (maximum score of 42) and the physical activity subscale (FABQpa) with 4 questions (maximum score of 24).
Return to work | between the end of the 2 weeks of initial treatment and 1 year of follow-up
  Number of days off work
Return to sport activities | between baseline and 1 year of follow-up
  Number of days off sports activities
Painful relapses | between baseline and 1 year of follow-up
  Number of new episodes of low back pain during follow-up. The patient indicates the start and end dates of each painful episode.
Analgesics consumption | over 12 months of follow-up
  The name of the treatment taken, the start and end dates and the doses of analgesics will be noted by the patient in the patient's diary.
Patient satisfaction regarding each program | one month of follow-up
  5-modality Likert scale developed specifically for the study

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Saint Martin, Pessac, France

IPD SHARING:
Plan to Share IPD: No